CLINICAL TRIAL: NCT01874184
Title: Diet, Exercise and Estrogen Metabolites Study (DEEM)
Brief Title: Group-Based Lifestyle Intervention in Measuring Biomarker Levels in Participants at High Risk for Breast Cancer
Acronym: DEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 9026; NCI-2014-00929 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 44358-J; 9026 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); R00NR012232 (NIH)
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Atypical Ductal Breast Hyperplasia; Atypical Lobular Breast Hyperplasia; BRCA1 Mutation Carrier; BRCA2 Mutation Carrier; Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (DEEM intervention) (Experimental): Participants take part in weekly 2-hour group counseling sessions for 6 months with taper beginning at 3 months. Group sessions include education, group process, and experiential learning on the benefits of physical activity, balanced nutrition, and mindfulness techniques. Participants set goals for changing their dietary habits with the help of a mental health counselor and are also encouraged to exercise 3-4 times per week, including experiential group activities such as brisk walking, yoga, Zumba, and group fitness.
  Interventions: Other: counseling intervention; Behavioral: behavioral dietary intervention; Behavioral: exercise intervention; Other: questionnaire administration; Other: laboratory biomarker analysis
- Arm II (usual care) (No Intervention): Participants receive their usual care and are provided with study materials on healthy diet and exercise at the end of the study.

INTERVENTIONS:
Other: counseling intervention — Take part in weekly group counseling sessions
  Other Names: counseling and communications studies
  Arms: Arm I (DEEM intervention)
Behavioral: behavioral dietary intervention — Set goals for changing dietary habits
  Arms: Arm I (DEEM intervention)
Behavioral: exercise intervention — Attend group exercise activities
  Arms: Arm I (DEEM intervention)
Other: questionnaire administration — Ancillary studies
  Arms: Arm I (DEEM intervention)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I (DEEM intervention)

SUMMARY:
This randomized clinical trial studies a group-based lifestyle intervention or usual care in measuring biomarker levels in participants at high risk for breast cancer. Studying the effects that changes to daily eating and exercise habits can have on the body's hormone levels and the body's ability to activate proteins may help doctors identify interventions for individuals at high risk for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To calculate eligibility rates, participation rates, retention, and adherence within the Diet, Exercise and Estrogen Metabolites (DEEM) study.

II. To determine inter- and intra-person variability of the estrogen-deoxyribonucleic acid (DNA) adducts (EDA) biomarkers in participants of the DFS.

III. To explore the effects of the intervention on percent adiposity and the EDA ratio at the end of the 3-month intervention and 6-month follow-up.

SECONDARY OBJECTIVES:

I. To explore the effects of the intervention on the DNA damage repair (DDR) biomarker at 3-months.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants take part in weekly 2-hour group counseling sessions for 6 months with taper beginning at 3 months. Group sessions include education, group process, and experiential learning on the benefits of physical activity, balanced nutrition, and mindfulness techniques. Participants set goals for changing their dietary habits with the help of a mental health counselor and are also encouraged to exercise 3-4 times per week, including experiential group activities such as brisk walking, yoga, Zumba, and group fitness.

ARM II: Participants receive their usual care and are also provided with study materials on healthy diet and exercise at the end of the study.

After completion of study, participants are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Women will be considered at high risk for developing breast cancer if they fulfill one of the following criteria:

  * A Gail model risk of >= 1.7% over 5
  * Claus model lifetime risk of > 20%
  * Tyrer-Cuzick model lifetime risk > 20%
  * Personal history of breast biopsy showing atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH) or lobular carcinoma in situ (LCIS)
  * Ductal carcinoma in situ (DCIS) that has been previously treated; patients must be at least 2 months from completion of primary therapy not currently on hormonal therapy
  * Deleterious mutation in breast cancer (BRCA)1 or BRCA2 another gene known to increase the risk of developing breast cancer
  * Risk assessment of 20% chance or greater of carrying a BRCA1/2 gene mutation; the BRCAPRO model will be used to assess this risk
* Body mass index (BMI)

  * For postmenopausal women: a BMI of > 28 and < 40
  * For premenopausal women: a BMI of > 25 and < 40
* Willingness to provide informed consent
* Physically able to undertake a moderate exercise program (assessed at the clinic visit)
* Participant has the ability to attend weekly group counseling sessions and subsequent clinic visits
* Participant has the ability to communicate in English
* Participant agrees to be randomly assigned

Exclusion Criteria:

* Women who are currently engaged in more than 90 min of moderate to vigorous exercise per week at the time of recruitment
* Alcohol/drug abuse or significant mental illness, as assessed by study personnel
* Previous diagnosis of invasive cancer within the past 5 years (in situ breast cancer and simple basal or squamous cell carcinoma not included)
* Plans to leave the geographic area within six months
* Contraindications for treadmill testing or entry into a training program
* Pregnant women or women planning to be pregnant in the following year will not be admitted in to the study

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Level of adherence to the dietary component evaluated using the 3-day food records | Up to 9 months
  Descriptive statistics will be calculated. The percentage of women meeting the study's eligibility criteria, percentage of those who agree to participate, and the percentage of those who complete the study will be stratified by intervention group. This analysis will summarize data collected from the participants' into themes.
Level of adherence to the exercise component evaluated using the physical activity logs | Up to 9 months
  Descriptive statistics will be calculated. The percentage of women meeting the study's eligibility criteria, percentage of those who agree to participate, and the percentage of those who complete the study will be stratified by intervention group. This analysis will summarize data collected from the participants' into themes.
Level of adherence to the group counseling sessions component evaluated by tracking attendance | Up to 9 months
  Descriptive statistics will be calculated. The percentage of women meeting the study's eligibility criteria, percentage of those who agree to participate, and the percentage of those who complete the study will be stratified by intervention group. This analysis will summarize data collected from the participants' into themes.
Inter-person variability | Up to 3 months
  The variance of the EDA biomarkers will be calculated in all participants at baseline, and stratify upon study arm. In order to determine the level of variance for biomarkers that is due to between-person variation in relation to the amount of variance that is due to within-person variance, the intra-class correlation coefficient will be calculated among the controls, which is based on the analysis of variance.
Change in EDA biomarker levels | Baseline to up to 6 months
  Linear regression models will be used for correlated outcomes.
Change in BMI | Baseline to up to 6 months
  Linear regression models will be used for correlated outcomes.
Change in percentage of total fat | Baseline to up to 6 months
  Linear regression models will be used for correlated outcomes.
Change in percentage of body fat as measured by BMI | Baseline to up to 6 months
  Linear regression models will be used for correlated outcomes.
Movement through the stages of change (pre-contemplation, contemplation, action, and maintenance) and data collected from quality of life questionnaires | Up to 9 months
  The participant's baseline level of readiness for change modified the effect of the intervention will be investigated, with the hypothesis that the largest impact will be observed within those with the highest level of readiness for change.

SECONDARY OUTCOMES:
Differences in change of the DNA repair assay in intervention participants versus controls | Baseline to up to 3 months
  Analysis of variance will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kerryn Reding, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Stone SA, Han CJ, Senn T, Korde LA, Allott K, Reding S, Whittington D, Reding KW. Sex Hormones in Women With Elevated Breast Cancer Risk Undergoing Weight Loss. West J Nurs Res. 2019 Nov;41(11):1602-1622. doi: 10.1177/0193945918820672. Epub 2019 Jan 7. PMID 30616442